CLINICAL TRIAL: NCT06932042
Title: Plant Dominant Low-protein Diet for Conservative Management of Chronic Kidney Disease: A Randomized Controlled Trial
Brief Title: PLADO for Conservative Management of CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese American University (Other)
Collaborators: Zayed University (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Rana Rizk, Assistant Professor, Lebanese American University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAU.SAS.RR4.2/Feb/2024
Record Dates: First submitted 2025-04-01; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease(CKD); Metabolic Acidosis
Keywords: Chronic kidney disease; metabolic acidosis; PLADO; Plant-dominant low protein diet; Nutrition education
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PLADO (Experimental)
  Interventions: Other: PLADO
- Standard-of-care diet (Active Comparator)
  Interventions: Other: Standard-of-care diet

INTERVENTIONS:
Other: PLADO — Low protein plant-dominant diet (PLADO) of 0.6-0.8 g/kg/day of proteins with at least 50% plant-based sources, sodium of <4 g/day and <3 g/day in case of edema or hypertension, fibers of 25-30 g/day, and calories of 30-35 Kcal/kg/day provided in the form of individualized meal plans administered by a licensed/registered dietitian. The nutrition education intervention will be provided via a primary face-to-face education/counseling session of 45-60 minutes, followed by a monthly face-to-face follow-up session of 30-45 minutes for 6 months, and a face-to-face follow-up session of 30-45 minutes after 3 months. At each visit, participants will be screened according to the Transtheoretical behavior change model (TTM) using a TTM-based algorithm to determine their stage/readiness to adhere to PLADO and will receive stage-based education and counseling accordingly. Stage-based education will be divided into 1) Pre-contemplation and contemplation; 2) Preparation; and 3) Action and Maintenance
  Arms: PLADO
Other: Standard-of-care diet — Current standard-of-care diet composed of dietary protein, fluid, sodium potassium, and phosphorus restrictions provided via monthly face-to-face sessions of 30-45 minutes over a period of 6 months, and a follow-up session after 3 months provided by the same licensed/registered dietitian. Patients will be recruited to the control arm in the same period to avoid seasonal differences.
  Arms: Standard-of-care diet

SUMMARY:
The goal of this clinical trial is to learn if a plant-dominant low protein diet, referred to as PLADO diet, works to decrease metabolic acidosis, a major risk factor for chronic kidney disease (CKD) progression, in adults with CKD. It will also learn about the safety, viability, and economic attractiveness of this diet.

The main questions it aims to answer are:

* Is the PLADO diet more effective in managing metabolic acidosis in comparison with the standard-of-care CKD diet in adults with CKD?
* Is the PLADO diet safe, viable, and economically attractive adults with CKD?

Researchers will compare the PLADO diet to the standard-of-care CKD diet to see if the PLADO diet works better to decrease metabolic acidosis.

Participants will:

* Receive nutrition education of the PLADO diet or the standard-of-care CKD diet via monthly sessions for 6 months.
* Visit the clinic monthly for 6 months, then after 3 months for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above, having controlled glycemic and blood pressure parameters on treatment, with an established diagnosis of stages 3-5 CKD and an estimated GFR ≤59 ml/min/1.73 m2 stable for at least three months, and with a normal nutritional status as defined by the GLIM criteria, attending the CKD outpatient clinics at LAUMC-RH, willing to undergo the baseline screening and attend the monthly face-to-face visits at the outpatient department at LAUMC-RH.

Exclusion Criteria:

* Patients with overt infection, persistent anorexia, vomiting, or diarrhea within the last month, presence of wasting diseases such as cancer, tuberculosis, liver failure, heart failure, and those with serum potassium >5.5 mEq/L during the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Metabolic acidosis assessed by PTCO2 | Baseline, Monthly for 6 months, Month 9

SECONDARY OUTCOMES:
Body weight | Baseline, Months 3, 6, and 9
  Body weight measured using a balance beam scale Unit: kg
%Weight Change | Months 3, 6, and 9
  %Weight Change (to the last measurement) Unit: %
Triceps Skinfold thickness | Baseline, Months 3, 6, and 9
  Triceps Skinfold thickness measured using a measuring tape and a skinfold caliper Unit: mm
Body Fat Percentage | Baseline, Months 3, 6, and 9
  %Body Fat for edema-free patients assessed using Bioimpedance analysis (Maltron Bioscan) Unit: %
Fat Free Mass Percentage | Baseline, Months 3, 6, and 9
  %Fat Free Mass for edema-free patients assessed using Bioimpedance analysis (Maltron Bioscan) Unit: %
Total Body Water Percentage | Baseline, Months 3, 6, and 9
  %Total Body Water for edema-free patients assessed using Bioimpedance analysis (Maltron Bioscan) Unit: %
Blood Urea Nitrogen (BUN) | Baseline, Monthly for 6 months, Month 9
  BUN assessed via blood test Unit: mg/dL
Estimated Glomerular Filtration Rate (eGFR) | Baseline, Monthly for 6 months, Month 9
  eGFR calculated using the Cockcroft-Gault equation = (((140 - age in years) x (weight in kg)) x 1.23) / (serum creatinine in micromol/l) Unit: mL/min/1.73m²
Serum Potassium (K) | Baseline, Monthly for 6 months, Month 9
  Serum K assessed via blood test Unit: mEq/L
Serum Phosphorus (P) | Baseline, Monthly for 6 months, Month 9
  Serum P assessed via blood test Unit: mg/dL
C-Reactive Protein (CRP) | Baseline, Months 3, 6, and 9
  Serum CRP assessed via blood test Unit: mg/L
Albumin | Baseline, Months 3, 6, and 9
  Serum Albumin assessed via blood test Unit: g/dL
Hemoglobin | Baseline, Months 3, 6, and 9
  Serum Hemoglobin assessed via blood test Unit: g/dL
Hematocrit | Baseline, Months 3, 6, and 9
  Serum Hematocrit assessed via blood test Unit: %
Mean Corpusculum Volume (MCV) | Baseline, Months 3, 6, and 9
  Average size of red blood cells assessed via blood test Unit: Femtoliter (fL)
Ferritin | Baseline, Months 3, 6, and 9
  Serum Ferritin assessed via blood test Unit: ng/mL
Glycated hemoglobin A1C | Baseline, Months 3, 6, and 9
  Glycated hemoglobin (A1C) measured via blood test Unit: %
Urinary microalbumin: creatinine ratio (UmACR) | Baseline, Months 3, 6, and 9
  UmACR assessed via urine test Unit: mg/g creatinine
Urinary potassium excretion | Baseline, Months 3, 6, and 9
  Urinary potassium excretion (spot) measured via urine test Unit: meq/L
Urinary phosphorus excretion | Baseline, Months 3, 6, and 9
  Urinary phosphorus excretion (spot) measured via urine test Unit: mg/dL
Global Leadership Initiative on Malnutrition (GLIM) criteria | Baseline, Months 3, 6, and 9
  GLIM criteria for the diagnosis of malnutrition. A participant is identified as malnourished when at least one phenotypic and one etiologic criterion is met. Phenotypic criteria include unintentional weight loss (>5% within 6 months or >10% beyond 6 months), age-specific low Body Mass Index (< 20 kg/m2 for individuals < 70 years old and < 22 kg/m2 for individuals 70 years and older), and reduced muscle mass assessed using body composition parameters to detect muscle depletion. Etiologic criteria include reduced food intake or assimilation (defined as a reduction in energy intake > 50% of requirements for over one week or any reduction lasting more than 2 weeks) and the presence of acute disease or chronic diseases related inflammation.
  Score: one phenotypic criterion and one etiologic criterion, to diagnose malnutrition
Total Caloric intake per kilogram body weight (Kcal/kg) | Baseline, Months 3, 6, and 9
  The total caloric intake will be assessed using a culturally specific quantitative Food Frequency Questionnaire (FFQ) crossed-checked with 24-hour recall series (one on a weekday and one on a weekend). The estimated total caloric intake (Kcal) will then be divided by the body weight (kg) at the same time point of data collection.
  Unit: Kcal/kg
Total dietary protein intake per kilogram body weight (g/kg) | Baseline, Months 3, 6, and 9
  The total dietary protein intake will be assessed using a culturally specific quantitative Food Frequency Questionnaire (FFQ) crossed-checked with 24-hour recall series (one on a weekday and one on a weekend). The estimated total amount of dietary proteins in grams (g) will then be divided by the dry body weight (kg) at the same time point of data collection.
  Unit: g/kg
Carbohydrate intake percentage (%) | Baseline, Months 3, 6, and 9
  The total carbohydrate intake will be assessed using a culturally specific quantitative Food Frequency Questionnaire (FFQ) crossed-checked with 24-hour recall series (one on a weekday and one on a weekend). The estimated total amount of carbohydrate in grams (g) will then be multiplied by 4 Kcal to get the calories of carbohydrates. Afterwards, it will be divided by the total amount of calories consumed at the same time point of data collection to obtain the percentage of total intake.
  Unit: percentage (%)
Total fat intake percentage (%) | Baseline, Months 3, 6, and 9
  The total fat intake will be assessed using a culturally specific quantitative Food Frequency Questionnaire (FFQ) crossed-checked with 24-hour recall series (one on a weekday and one on a weekend). The estimated total amount of fat in grams (g) will then be multiplied by 9 Kcal to get the calories of fat. Afterwards, it will be divided by the total amount of calories consumed at the same time point of data collection to obtain the percentage of total intake.
  Unit: percentage (%)
Trans fat intake percentage (%) | Baseline, Months 3, 6, and 9
  The total trans-fat intake will be assessed using a culturally specific quantitative Food Frequency Questionnaire (FFQ) crossed-checked with 24-hour recall series (one on a weekday and one on a weekend). The estimated total amount of trans-fat in grams (g) will then be multiplied by 9 Kcal to get the calories of fat. Afterwards, it will be divided by the total amount of calories consumed at the same time point of data collection to obtain the percentage of total intake.
  Unit: percentage (%)
Total potassium intake (g) | Baseline, Months 3, 6, and 9
  The total potassium intake will be assessed using a culturally specific quantitative Food Frequency Questionnaire (FFQ) crossed-checked with 24-hour recall series (one on a weekday and one on a weekend) and reported in grams per day.
  Unit: g/d
Total phosphorus intake (g) | Baseline, Months 3, 6, and 9
  The total phosphorus intake will be assessed using a culturally specific quantitative Food Frequency Questionnaire (FFQ) crossed-checked with 24-hour recall series (one on a weekday and one on a weekend) and reported in grams per day.
  Unit: g/d
Total sodium intake (g) | Baseline, Months 3, 6, and 9
  The total sodium intake will be assessed using a culturally specific quantitative Food Frequency Questionnaire (FFQ) crossed-checked with 24-hour recall series (one on a weekday and one on a weekend) and reported in grams per day.
  Unit: g/d
Nutrition focused physical examination (NFPE) | Baseline, Months 3, 6, and 9
  The nutrition focused physical examination will be conducted by a licensed dietitian who will assess fat and muscle depletion, as well as the presence of edema.
Muscle strength (kg) | Baseline, Months 3, 6, and 9
  Muscle strength will be measured using a handgrip strength assessment with a calibrated hand dynamometer. Participants will be seated upright with their back supported, feet flat on the floor, and their elbow flexed at a 90-degree angle. The hand dynamometer will be adjusted to fit the participant's hand size who will be instructed to squeeze the dynamometer with maximum effort for 3-5 seconds. Three measurements will be taken for each hand, with a rest period of 30 to 60 seconds and the average of the three measurements will be recorded as the final handgrip strength.
  Unit: kg
Gastrointestinal Symptoms | Baseline, Monthly for 6 months, Month 9
  Gastrointestinal symptoms will be assessed using the Birmingham IBS Symptom Questionnaire (B-IBS-Q), a validated tool for evaluating the frequency, severity, and impact of gastrointestinal symptoms. It is a self-administered questionnaire consisting of 11 items designed to assess the frequency of IBS-related symptoms, with each question having a standard response scale. Symptoms are measured based on a 6-point Likert scale (0-5) ranging from all of the time (5) to none (0) and converted to 100, with higher scores indicating more frequent IBS symptoms. The scale has 3 dimensions, including pain, constipation, and diarrhea.
Health-related Quality of Life | Baseline, Months 3, 6, and 9
  Quality of life will be assessed using the EuroQOL-5D-5L (EQ-5D-5L), a widely validated and internationally recognized instrument for measuring health-related quality of life. The tool consists of two components: a descriptive system and a visual analog scale (VAS). The descriptive component includes five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 5-level scale, ranging from no problems to extreme problems. Participants will select the most appropriate level that reflects their current health status for each dimension. The responses are then used to generate a health state profile, which can be converted into a single index score using country-specific value sets. In addition to the descriptive system, participants will rate their overall health status using a visual analog scale (VAS), ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Costs | Baseline, Months 3, 6, and 9
  Costs relevant to direct medical costs, direct non-medical costs, and indirect costs assessed using a resource utilization questionnaire with the patients, and calculated following the identification, measurement, and valuation steps.

CONTACTS AND LOCATIONS:
Locations (1):
- Lebanese American University Medical Center- Rizk Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No